CLINICAL TRIAL: NCT00629499
Title: Phase II Trial of Nanoparticle Albumin-Bound (Nab) Paclitaxel/Cyclophosphamide in Early-Stage Breast Cancer (With Trastuzumab in HER2 Positive Patients)
Brief Title: Nanoparticle Albumin-Bound (Nab) Paclitaxel/Cyclophosphamide in Early-Stage Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 116
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Results first posted 2012-12-20 (Estimated); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
Keywords: Early Stage Breast Cancer; Her2-positive; nab paclitaxel; cyclophosphamide; trastuzumab
MeSH Terms: conditions — Breast Neoplasms | interventions — Taxes; Albumin-Bound Paclitaxel; Cyclophosphamide; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): 100 mg/m2 of intravenous (IV) nab paclitaxel weekly (i.e., on Days 1, 8, and 15 of each 3 week treatment cycle) in combination with 600 mg/m2 of IV cyclophosphamide once every 3 weeks for 4 cycles (i.e., a total treatment period of 12 weeks [84 days]). Patients with fluorescence in situ hybridization (FISH) HER2+ or IHC3+ breast cancer will also receive treatment with trastuzumab in addition to the nab paclitaxel / cyclophosphamide combination therapy. Maintenance therapy with trastuzumab will continue (for the HER2+ patients who are receiving trastuzumab) after the 12-week treatment period with combination nab paclitaxel/cyclophosphamide/trastuzumab. The total treatment time for trastuzumab will be 52 weeks rather than only 12 weeks.
  Interventions: Drug: nab paclitaxel; Drug: Cyclophosphamide; Drug: Trastuzumab

INTERVENTIONS:
Drug: nab paclitaxel — 100 mg/m2 of intravenous (IV) nab paclitaxel weekly (i.e., on Days 1, 8, and 15 of each 3 week treatment cycle)
  Other Names: Abraxane
Drug: Cyclophosphamide — 600 mg/m2 of IV cyclophosphamide
  Other Names: Cytoxan
Drug: Trastuzumab — 8 mg/kg loading dose of IV trastuzumab will be administered on Day 1, followed by doses of 6 mg/kg IV trastuzumab once every 3 weeks.
  Other Names: Herceptin

SUMMARY:
This is a non-randomized, Phase II study. Efficacy is not a primary endpoint in this study; however, progression-free survival will be followed and determined for the patients in this study. Approximately 50 patients are planned to be enrolled in this study.

DETAILED DESCRIPTION:
Given the favorable activity demonstrated in a trial using the taxane docetaxel in combination with cyclophosphamide, we propose a Phase II trial of 4 cycles of weekly nab paclitaxel combined with cyclophosphamide. The favorable toxicity profile for weekly nab paclitaxel, in addition to its demonstrated superiority over standard paclitaxel in early-stage breast cancer, makes it an ideal taxane to evaluate in this setting. In this study, nab paclitaxel will be administered once weekly, in combination with q3wk cyclophosphamide. By using this combination therapy method, the goal of this study is to maximize the opportunity to demonstrate improved tolerability of adjuvant nab paclitaxel using a weekly dosing schedule in combination with q3wk cyclophosphamide.

In this study, patients who demonstrate FISH or IHC3+ HER2 positivity and adequate cardiac function will also receive treatment with trastuzumab in addition to the nab paclitaxel / cyclophosphamide combination therapy. Trastuzumab will be administered IV using an 8 mg/kg loading dose on Day 1 of the treatment period. If no toxicity occurs, subsequent doses of trastuzumab will be administered IV as a 6 mg/kg dose approximately every 21 days for a total of 52 weeks (thus, maintenance therapy with trastuzumab will continue after the 12-week period of combination therapy with nab paclitaxel/cyclophosphamide/trastuzumab has ended).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive adenocarcinoma of the breast or inflammatory breast cancer, with an interval between definitive breast surgery and study registration of <60 days.
* Definitive surgical treatment must be either mastectomy or breast-conserving therapy with axillary lymph node dissection for operable breast cancer (pT1 4 [including inflammatory breast cancer], pN0 3, and M0). Margins of resected specimen from definitive surgery must be histologically free of invasive adenocarcinoma and ductal carcinoma in situ (DCIS). Lobular carcinoma in-situ does not count as a positive margin.
* Patients with ≥1 axillary lymph node containing metastatic adenocarcinoma measuring >0.2 mm, OR lymph node-negative patients with high-risk features
* Patients with HER2/neu positive or negative tumors (HER2 positivity must be documented by FISH positivity or IHC 3+).
* Patients who are to receive trastuzumab must have normal cardiac function (MUGA [cardiac ejection fraction >50%, or greater than or equal to the institutional lower limit of normal], or echocardiogram [ECHO] within institutional normal limits).
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤2.
* Patients who are either chemotherapy naïve, or who have received prior chemotherapy >5 years ago.
* Patients with previous invasive cancers (including breast cancer) eligible only if treated >5 years prior to entering this study, and show no evidence of recurrent disease.
* Adequate bone marrow function
* Adequate liver function,
* Adequate renal function,
* Patients of childbearing potential must use an effective method of contraception that is acceptable to their study physician from the time of signing informed consent until at least 3 months after the last dose of protocol treatment, and must have a negative pre study serum pregnancy test.
* Pre-existing peripheral neuropathy must be less than or equal to grade 1 by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0 criteria.
* MammoSite® brachytherapy radiation accepted when performed immediately following surgery and prior to receiving chemotherapy.
* Patients with bilateral, synchronous breast cancer, provided that one primary tumor meets the inclusion criteria.

Exclusion Criteria:

* Patients who are pregnant or breastfeeding.
* M1 metastatic disease.
* Patients requiring neoadjuvant chemotherapy.
* Life expectancy of greater than 6 months.
* History of cardiac disease, with a New York Heart Association (NYHA) Class II or greater CHF
* Myocardial infarction (MI) or unstable angina in the past 12 months prior to Day 1 of treatment, serious arrhythmias requiring medication for treatment, any history of stroke or transient ischemic attack at any time, clinically significant peripheral vascular disease, or evidence of a bleeding diathesis or coagulopathy.
* Any investigational agent within 30 days of receiving the first dose of study drug.
* Treatment with prior trastuzumab or bevacizumab therapy.
* Concurrent treatment with any other anti-cancer therapy is not permitted.
* History of significant psychiatric disorders.
* History of active, uncontrolled infection.
* A serious, non-healing wound, ulcer, or bone fracture.
* Any other diseases, metabolic dysfunction, findings from a physical examination, or clinical laboratory test results that give reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, that may affect the interpretation of the results or that renders the patient at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Hainsworth, MD, Study Chair — SCRI Development Innovations, LLC
Locations (10):
- United States (10):
  - Watson Clinic Center for Cancer Care and Research, Lakeland, Florida
  - Gulfcoast Oncology Associates, St. Petersburg, Florida
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Mercy Hospital, Portland, Maine
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - St. Louis Cancer Care, Chesterfield, Missouri
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Peninsula Cancer Institute, Newport News, Virginia

REFERENCES:
- [Result] Yardley D, Burris H 3rd, Peacock N, Raefsky E, Melnik M, Inhorn R, Shipley D, Hainsworth J. A pilot study of adjuvant nanoparticle albumin-bound (nab) paclitaxel and cyclophosphamide, with trastuzumab in HER2-positive patients, in the treatment of early-stage breast cancer. Breast Cancer Res Treat. 2010 Sep;123(2):471-5. doi: 10.1007/s10549-010-1047-0. Epub 2010 Jul 24. PMID 20658263
- See also: PubMed — http://www.ncbi.nlm.nih.gov/pubmed/20658263

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 63
Completed | 63
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 63
Age, Continuous [Median (Full Range); unit: years] | 57 [27 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Remained Alive Without Evidence of Recurrence as a Measure of Tolerability of Adjuvant Nab Paclitaxel
Time Frame: 18 Months
Population: Patients were analyzed if they remained alive and without evidence of recurrence.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 63
Participants | 63

2. Secondary Outcome: Disease-free Survival
Description: Number of participants that are disease free at 18th month
Time Frame: 18 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 63
Participants | 63

3. Secondary Outcome: Overall Survival
Description: Number of participants that are alive at 18th month
Time Frame: 18 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 63
Participants | 63

ADVERSE EVENTS:
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 4/63
Other Adverse Events (participants affected / at risk) | 59/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=63)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient fell down flight of stairs causing multiple fractures. Event unrelated to protocol therapy.
Mental Status (Nervous system disorders) | 1 (1)
Hemorrhage - GI (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=63)
Hemoglobin (Blood and lymphatic system disorders) | 14 (14) — Anemia
Neutrophils (Blood and lymphatic system disorders) | 48 (48) — Neutropenia
Fatigue (General disorders) | 26 (26)
Nausea (Gastrointestinal disorders) | 14 (14)
Arthralgia/Myalgia (Musculoskeletal and connective tissue disorders) | 21 (21)
Rash (Skin and subcutaneous tissue disorders) | 8 (8)
Vomiting (Gastrointestinal disorders) | 7 (7)
Neuropathy (Nervous system disorders) | 5 (5) — Peripheral Neuropathy
Diarrhea (Gastrointestinal disorders) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 31 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.